CLINICAL TRIAL: NCT04258033
Title: A Phase II, Open-label, Multicenter and Multi-cohorts Study to Evaluate the Efficacy and Safety of PLB1001 in Advanced Non-small Cell Lung Cancer With c-Met Dysregulation
Brief Title: A Study of PLB1001 in Non-small Cell Lung Cancer With c-Met Dysregulation(KUNPENG)
Acronym: KUNPENG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001-II-NSCLC-01
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLB1001 (Experimental): Subjects will receive 200mg of PLB1001 twice daily in cycles of 28-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: PLB1001

INTERVENTIONS:
Drug: PLB1001 — PLB1001 is a capsule in the form of 25 mg and 100mg, twice daily.
  Other Names: Bozitinib

SUMMARY:
This is a Phase II, open-label, multicenter and multi-cohorts study of PLB1001 administered orally twice daily to locally advanced/metastatic NSCLC patients with c-Met dysregulation.

DETAILED DESCRIPTION:
PLB1001 will be administrated 200mg twice daily. The treatment will be discontinued for the patients who experience disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent. A cycle of study treatment will be defined as 28 days of continuous dosing. The study includes 4 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Histologically or cytologically confirmed advanced non-small cell lung cancer
* Must have evidence of c-Met dysregulation from the results of molecular pre-screening evaluations
* At least one measurable lesion as per RECIST v1.1
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1
* ECOG Performance Status of 0-1.

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases that are neurologically unstable or requiring increasing doses of steroids to control, and patients with any CNS deficits.
* Clinically significant, uncontrolled heart diseases Unstable angina History of documented congestive heart failure (New York Heart Association functional classification > II) Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg Arrhythmias
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
* Major surgery within 4 weeks prior to starting PLB1001
* Previous anti-cancer and investigational agents within 2 weeks before first dose of PLB1001. If previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 4 weeks before first dose of PLB1001
* Pregnant or nursing women
* Involved in other clinical trials < 2 weeks prior to Day. If previous treatment of clinical trial is a monoclonal antibody, then the treatment must be discontinued at least 4 weeks before first dose of PLB1001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  Objective response rate will be determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Objective response rate is defined as the percentage of patients who experienced either a complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Progression free survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause. PD is defined as at least a 20 % increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Overall survival | 4 years
  Overall survival is defined as the time (in months) from first trial treatment administration to the date of death.
Disease control rate | 2 years
  Disease control rate according to RECIST 1.1 is the percentage of patients who experienced either a complete response (CR), partial response (PR) or stable disease (SD).
Time to response | 2 years
  Time to response according to RECIST 1.1 is the time from the first trial treatment administration to the CR/PR (whichever is first) criteria are first met. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Duration of response | 2 years
  Duration of response according to RECIST 1.1 is the time from when the CR/PR (whichever is first) criteria are first met until progression of disease (PD) or death due to any cause. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Occurrence of Treatment emergent adverse event (TEAEs) | 2 years
  This outcome measure will be presented as the percentage of subjects with any (serious) adverse event (AE). Percentages are calculated using total number of subjects per treatment cohort as the denominator.
Maximum Plasma concentration (Cmax) of drug | Cycle 1, Day 1 and on Cycle 1, Day 15
  In the study some Pharmacokinetics (PK) profiles of PLB1001 will be obtained following administration of PLB-1001 at pre-dose and at the 0.5, 2, 4, 6,10 hours time points on Cycle 1, Day 1 and on Cycle 1, Day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu YL, Yao Y, Yang JJ, Wu L, Zhang W, Wang Y, Xu HP, Song Y, Zhang Y, Zhao J, Chen JH, Wang ZH, Wang QM, Hu J, Li XY, Fan Y, Chen Y, Fang J, Han D, Xue WZ, Liu SM, Zhou Q, Zhang PL, Shi HP. Vebreltinib in MET amplification-driven advanced non-small-cell lung cancer (KUNPENG): a single-arm, multi-cohort, multicentre, phase 2 study. Lancet Oncol. 2026 Jan;27(1):36-44. doi: 10.1016/S1470-2045(25)00594-7. Epub 2025 Dec 6. PMID 41365311
- [Derived] Yang JJ, Zhang Y, Wu L, Hu J, Wang ZH, Chen JH, Fan Y, Lin G, Wang QM, Yao Y, Zhao J, Chen Y, Fang J, Song Y, Zhang W, Cheng Y, Guo RH, Li XY, Shi HP, Xue WZ, Han D, Zhang PL, Wu YL. Vebreltinib for Advanced Non-Small Cell Lung Cancer Harboring c-Met Exon 14 Skipping Mutation: A Multicenter, Single-Arm, Phase II KUNPENG Study. J Clin Oncol. 2024 Nov;42(31):3680-3691. doi: 10.1200/JCO.23.02363. Epub 2024 Jul 26. PMID 39058972
- [Derived] Huang S, Li L, Yan N, Zhang H, Guo Q, Guo S, Geng D, Liu X, Li X. Case report: The effect of second-line vebreltinib treatment on a patient with advanced NSCLC harboring the MET exon 14 skipping mutation after tepotinib treatment. Front Oncol. 2024 Apr 19;14:1331387. doi: 10.3389/fonc.2024.1331387. eCollection 2024. PMID 38706592